CLINICAL TRIAL: NCT03120507
Title: Resuscitation Outcomes in the Netherlands Study
Brief Title: Resuscitation Outcomes in the Netherlands
Acronym: ROUTiNE
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Marc Schluep, Principal Investigator, Erasmus Medical Center
Other Study IDs: ABR55661.078.16; NTR6145 (Other: Dutch Trial Registry); MEC-2016-563 (Other: Erasmus MC METC)
Record Dates: First submitted 2017-04-06; First posted 2017-04-19 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Heart Arrest; Cardiac Arrest; Cardiac Arrest as A Complication of Care; Outcome, Fatal; Quality of Life; Cognitive Impairment
Keywords: in-hospital cardiac arrest; IHCA; quality of life; QoL; patient-reported outcomes
MeSH Terms: conditions — Heart Arrest; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Resuscitation Outcomes in the Netherlands - study assesses one-year survival and quality of life after In-Hospital Cardiac Arrest(IHCA). It's design is a multicenter prospective observational cohort study which will include all patients undergoing cardiopulmonary resuscitation (CPR) for IHCA in 2017. Current literature describes poor survival after IHCA and no risk stratification tool for long-term outcome is available. Furthermore no such study has ever been performed in the Netherlands. The investigators aim to gain further insight in this major adverse event.

DETAILED DESCRIPTION:
Background: In-hospital cardiac arrest (IHCA) is a serious adverse event for which cardiopulmonary resuscitation (CPR) can be performed to restore circulation. Currently survival after IHCA is poor. To assess the success of resuscitation attempts there is a need for research that focuses on long-term survival and quality of life. Patient selection for CPR, prevention of cardiac arrest and improvement of CPR techniques are crucial for improving qualitative survival. To assess the feasibility of this project a single-center retrospective cohort study was conducted over a 10-year period in the OLVG hospital. For all patients who received CPR survival to discharge was 32% and one-year survival was 22%. This is slightly higher than survival reported in contemporary literature. Due to it's design no prognostic variables could be derived from this study, however data suggested age and Charlson Comorbidity Index could prove useful in predicting long-term outcome. In the consecutive year this study was designed.

Hypothesis: The hypothesis is that one-year survival after IHCA in Dutch hospitals is poor, consistent with international literature and our feasibility trial, and survival can be improved through selection, prevention and training.

Objective: The main objective of this study is to assess the one-year survival of patients after CPR for in-hospital cardiac arrest. The secondary objectives are to assess quality of life and functional status after successful CPR. Furthermore the investigators aim to assess if there are patient-related predicting factors for these outcome measures and to assess whether outcomes are influenced by hospital-related factors (i.e. CPR training and treatment options).

Study design: The current study has a prospective, observational design, with a 12-month follow-up. Patients will be included from January 1st 2017. Patient data collection will take place at four time points: T0= directly post-CPR, T1= at hospital discharge or at in-hospital death, T2= 3 months after CPR, T3= 12 months after CPR. Clinical data will be collected at all time points. Quality of life data will be collected at T2 and T3 by means of validated questionnaires. We will assess functional status through questionnaires and link these to pre-existing and acquired comorbidities (e.g. stroke). General hospital data and data concerning the level of CPR-training will be ascertained at four moments during the first year of patient inclusion.

Study population: An estimated six hundred patients of 18 years or older who will receive CPR for cardiac arrest in the participating hospitals. This will include all cases of in-hospital cardiac arrest, also including Operation Room (OR), Intensive/Coronary Care Unit (ICU/CCU) and Emergency Department (ER). Patients in whom CPR was started before arrival in hospital will be excluded.

Expected results: The main study endpoints are one-year survival and quality of life. Secondary endpoints are direct survival and survival to discharge. The first preliminary results are expected in the first quarter of 2018. After conclusion of this project the investigators of this project aim to develop recommendations that will improve survival after IHCA.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Receiving cardiopulmonary resuscitation, as defined by starting manual chest compressions, for a circulatory arrest occuring in-hospital.
* In hospital is defined as all hospital wards, departments, outpatient clinics, and hallways.

Exclusion Criteria:

* Children (<18 years of age)
* Purposely induced cardiac arrest (e.g. cardiac surgery)
* Purposely induced arrhythmias (e.g. electrophysiological treatment)
* Refusal to participate
* Primary out-of-hospital cardiac arrest with re-arrest <24h after hospital admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: An estimated six hundred patients of 18 years or older who will receive CPR for cardiac arrest in the participating hospitals (n=15). This will include all cases of in-hospital cardiac arrest, also including Operation Room (OR), Intensive/Coronary Care Unit (ICU/CCU) and Emergency Department (ER). Patients in whom CPR was started before arrival in hospital will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
one-year survival | one year
  Survival one year after in-hospital cardiac arrest

SECONDARY OUTCOMES:
SF-12 | 3 months and one year after in-hospital cardiac arrest
  Quality of life measured by SF-12 questionnaire
EuroQoL | 3 months and one year after in-hospital cardiac arrest
  Quality of life measured by EuroQoL questionnaire
HADS | 3 months and one year after in-hospital cardiac arrest
  Quality of life measured by Hospital Anxiety and Depression Scale questionnaire
Charlson Comorbidity Index | 3 months and one year after in-hospital cardiac arrest
  Development of new comorbidities as defined by the Charlson Comorbidity Index.
Cardiovascular events | 3 months and one year after in-hospital cardiac arrest
  Development of new cardiovascular events (e.g. myocardial infarction, stroke), by means of checkbox question.
Working life | Prior to in-hospital cardiac arrest and 3 months and one year after in-hospital cardiac arrest
  Participation in working life; status before cardiac arrest and after by means of checkbox question.
TICS | 3 months after in-hospital cardiac arrest, if patients are not able to respond to regular questionnaires (paper)
  Telephonic interview for Cognitive Status
CSI | 3 months and one year after in-hospital cardiac arrest
  Caregiver strain index for caregivers of In-Hospital Cardiac Arrest Survivors

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jan Stolker, MD PhD, Principal Investigator — Erasmus Medical Center; Marc Schluep, MD, Principal Investigator — Erasmus Medical Center; Sanne Hoeks, PhD, Study Chair — Erasmus Medical Center; Henrik Endeman, MD PhD, Study Chair — OLVG
Locations (12):
- Netherlands (12):
  - Rijnstate Ziekenhuis, Arnhem, Gelderland
  - OLVG, Amsterdam, North Holland
  - Deventer Ziekenhuis, Deventer, Overijssel
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Isala klinieken, Zwolle, Overijssel
  - Amphia Ziekenhuis, Breda, South Holland
  - Reinier de Graaf Gasthuis, Delft, South Holland
  - Albert Schweitzer Ziekenhuis, Dordrecht, South Holland
  - Sint Franciscus Vlietland Groep, Rotterdam, South Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - Haaglanden Medisch Centrum, The Hague, South Holland
  - ZorgSaam Zeeuws-Vlaanderen, Terneuzen, Zeeland

IPD SHARING:
Plan to Share IPD: No